CLINICAL TRIAL: NCT03036306
Title: A Randomized, Placebo Controlled, Double-blind, Dose Ranging Study to Evaluate the Safety and Tolerability of SCX-001 Cream in Healthy Volunteers With Induced Dermal Incisions
Brief Title: Dose Ranging Study to Evaluate the Safety and Tolerability of SCX-001 Cream in Healthy Volunteers With Induced Dermal Incisions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ScarX Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCX-001-1
Record Dates: First submitted 2017-01-16; First posted 2017-01-30 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Scarring
Keywords: scar; nefopam; cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.0 % SCX-001 cream (Experimental): Subjects randomized to this arm will have one lateral hip wound treated with 1.0% SCX-001 cream and one wound treated with placebo. Intra-subject hip wound treatment is randomly allocated
  Interventions: Drug: SCX-001
- 3.0% SCX-001 cream (Experimental): Subjects randomized to this arm will have one lateral hip wound treated with 3.0% SCX-001 cream and one wound treated with placebo. Intra-subject hip wound treatment is randomly allocated
  Interventions: Drug: SCX-001
- Placebo cream (Placebo Comparator): Subjects randomized to this arm will have both lateral hip wounds treated with Placebo cream. Intra-subject hip wound treatment is randomly allocated
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SCX-001 — Nefopam cream formulation
  Arms: 1.0 % SCX-001 cream; 3.0% SCX-001 cream
Other: Placebo — Cream formulation without Nefopam
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to assess the safety and local tolerability of two different concentrations of of SCX-001 cream, as compared to placebo, when topically applied twice a day for 21 days to artificially induced dermal wounds in healthy volunteers. In addition, the absorption and elimination of profiles of this topically applied product will be determined through pharmacokinetic sampling. Assessments for effect of SCX-001 vs. placebo will be done but are considered exploratory.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged ≥18 - ≤65 years who have voluntarily signed and dated an Informed Consent Form (ICF).
2. Subjects with, in the opinion of the Investigator, clinically acceptable results at screening for the laboratory tests specified in the trial protocol.
3. Women of child bearing potential must provide a negative pregnancy serum/urine test at time of screening and have to be compliant with an effective form of birth control throughout the entire study.* Non-child bearing potential means subjects have had a history of tubal ligation or a hysterectomy or are post-menopausal with no menses for at least 1 year prior to enrolment in the study.
4. Subjects, who are, in the opinion of the Investigator, able to understand the study, co- operate with the study procedures and are willing to return to the clinic for all of the required follow-up visits.
5. Subjects must be able to cooperate with requirements of the study (e.g. able to speak, read and write English, expect to be available for adverse event monitoring for the duration of the study).

Exclusion Criteria:

1. Subjects who have scarring from previous interventions or evidence of thermal, electrical or radiation burn scars, tattoos, birthmarks or moles within 5 cm of the treatment site.
2. Subjects with a history or family history of keloid formation.
3. Subjects with a concurrent illness or condition that may have interfered with wound healing like neoplastic, immune-mediated, or primary infectious disease (e.g. carcinoma, vasculitis, connective tissue disease, immune system disorders, rheumatoid arthritis, chronic renal impairment, significant hepatic impairment, inadequately or uncontrolled congestive heart failure or diabetes mellitus) or any clinically significant medical condition or history of any condition which may impair wound healing.
4. Subjects with a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of acute wounds or will involve the areas to be examined in this trial (including psoriasis, dermatitis, eczema)
5. Subjects with a body mass index <15 or >35 kg/m2.
6. A history of radiotherapy to the study scar area.
7. Subjects who have used nicotine-containing products (including vaping) within one month prior to the screening visit.
8. Subjects who are positive for HIV, hepatitis B or C.
9. Subjects who have known sensitivities to SCX-001 Cream, structurally related compounds or any of the constituents of SCX-001 Cream.
10. Subjects who have known sensitivities to EMLA cream, chlorhexidine or adhesive dressings
11. Subjects with a history of any malignancy in the five years prior to the screening visit.
12. Subjects with a life expectancy of <9 months, terminal conditions or factors making follow-up difficult (e.g. no fixed address, telephone etc.).
13. Subjects with planned major surgical intervention during the course of the study.
14. Subjects who have received corticosteroids, immunosuppressive agents, anticoagulants, radiation therapy or chemotherapy at a dose that might have interfered with wound healing within the last 90 days prior to study enrolment.
15. Subjects who have received NSAIDS or ASA in the past week.
16. Subjects with a creatinine clearance of 80 ml/min or less.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01; Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events and Tolerability Assessments | 4 months
  Adverse events, Tolerability assessments

SECONDARY OUTCOMES:
Scar Size | 4 months
  Repeat measurement of scar size by ultrasound following wound closure to the end of study and digital camera following wounding to the end of the study
Scar Quality | 4 months
  Repeat measurement of erythema and pigmentation of scars by mexameter following wound closure to the end of study
Time to Wound Closure | 4 months
  Repeat examination of wounds for closure defined as 100% epithelialization of the wound with no exudate observed assessed form time of wounding to wound closure on both hips
Area under the plasma concentration-time curve (AUC) | 4 weeks
  Serial serum samples to determine AUC (0-6h, 0-8h)
Time to reach maximum observed plasma concentration (Tmax) | 4 weeks
  Serial serum samples to determine Tmax
Maximum observed plasma concentration (Cmax) | 4 weeks
  Serial serum samples to determine Cmax
Gene expression analysis | Done on the day of the last dose of treatment (20 days following wounding)
  RT-qPCR on scar biopsy samples
Histological analysis | Done on the day of the last dose of treatment (20 days following wounding)
  Immunohistochemistry on scar biopsy samples
Collagen orientation analysis | Done on the day of the last dose of treatment (20 days following wounding)
  Collagen orientation index on scar biopsy samples
Overall Satisfaction | 4 months
  Repeat measurement of both subject and investigator satisfaction with scar appearance by Subject and Observer Scar Assessment Scale (POSAS) following wound closure to the end of study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No